CLINICAL TRIAL: NCT03096730
Title: The Effect of Dexmedetomidine Combined With Low-dose Nalmefene on Preventing Remifentanil-induced Postoperative Hyperalgesia in Patients Undergoing Gynecological Surgery
Brief Title: Effect of Dexmedetomidine Combined With Low-dose Nalmefene on Preventing Remifentanil-induced Postoperative Hyperalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang003
Record Dates: First submitted 2017-03-13; First posted 2017-03-30 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Pain; Anesthesia
Keywords: Remifentanil; Opioid-induced hyperalgesia; Postoperative pain; pain intensity
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Saline Solution; Sodium Chloride; Remifentanil; Injections; Sufentanil; Dexmedetomidine; nalmefene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Normal Saline (Placebo Comparator): Normal saline is intravenously administrated before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Normal saline; Drug: Remifentanil
- Sufentanil (Sham Comparator): Normal saline is intravenously admistrated before anesthesia induction and intraoperative pain management was with sufentanil
  Interventions: Drug: Normal saline; Drug: Sufentanil
- Dexmedetomidine (Active Comparator): Dexmedetomidine is intravenously administrated at a dose of 0.5ug/kg 10min before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine injection
- Nalmefene (Active Comparator): Nalmefene is intravenously administrated at a dose of 0.2ug/kg before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Remifentanil; Drug: Nalmefene
- Dexmedetomidine-Nalmefene (Active Comparator): A dose of 0.1ug/kg nalmefene and a dose of 0.25ug/kg dexmedetomidine for 10 minutes before anesthesia induction and intraoperative pain management was with remifentanil
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine injection; Drug: Nalmefene

INTERVENTIONS:
Drug: Normal saline — Normal saline is intravenously administrated before anesthesia induction
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal Saline; Sufentanil
Drug: Remifentanil — Remifentanil is intravenously administrated
  Other Names: Remifentanil Hydrochloride for Injection
  Arms: Dexmedetomidine; Dexmedetomidine-Nalmefene; Nalmefene; Normal Saline
Drug: Sufentanil — Sufentanil is intravenously administrated
  Other Names: Sufentanil injection
  Arms: Sufentanil
Drug: Dexmedetomidine injection — Dexmedetomidine is intravenously administrated before anesthesia induction
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine; Dexmedetomidine-Nalmefene
Drug: Nalmefene — Nalmefene is intravenously administrated before anesthesia induction
  Arms: Dexmedetomidine-Nalmefene; Nalmefene

SUMMARY:
To explore and compare antihyperalgesic effects of Dexmedetomidine,Nalmefene,and a combination of both received before anesthesia induction.

To evaluate and examine the incidence of adverse effects with the purpose of selecting the optimum dose.

DETAILED DESCRIPTION:
There are a dramatically increasing number of evidences that administration of the potent, ultra-short-acting opioid remifentanil seems to cause opioid-induced hyperalgesia (OIH) more frequently and predictably compared with the others, likely due to its rapid onset and offset. Therefore, prophylaxis of remifentanil induced hyperalgesia is indispensable to postoperative comfort and satisfaction.

There is no denying the fact that OIH is related to central glutaminergic system and N-methyl-d-aspartate(NMDA)receptor-activation induced central sensitization. Dexmedetomidine is an 2-adrenergic agonist that has been shown to synergize with opioids. Dexmedetomidine inhibits NMDAR excitability by reducing the phosphorylation of N-methyl-D-aspartate receptor 2B subunit phosphorylation of spinal dorsal horn induced by remifentanil, thereby achieving the goal of reducing OIH. Nalmefene is a pure opioid receptor antagonist that antagonizes the Mu receptor, alleviating the central sensitization of NMDA, thereby reducing OIH. At the same time reported in the literature, opioid receptor has a bimode：On the one hand can be mediated by Gs protein-mediated pain, respiratory depression, nausea and vomiting, etc ; on the other hand can be coupled with Gi / Go protein mediated analgesic effect. Low-dose nalmefene (<1.0ug / kg) and other opioid receptor antagonists can antagonize the role of Gs protein-coupled opioid receptors, blocking the pathway of opioid excitatory effects, thereby reducing the incidence of adverse reactions.The following study is carried out to evaluate whether dexmedetomidine combined with nalmefene can be safely and effectively applied to prevent postoperative hyperalgesia induced by remifentanil in patients undergoing Laparoscopic gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are scheduled to undergo Gynecological surgery under a short general anesthesia of 1-3 hours.
2. American Society of Anesthesiologists physical status is I-II.
3. Written informed consent was obtained from all the subjects.

Exclusion Criteria:

1. Subject has a diagnosis of Coronary heart disease, bronchial asthma, cardiac, lung, hepatic and renal insufficiency.
2. Subject has a diagnosis of Severe high blood pressure , diabetes, obesity (BMI>30).
3. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre-existing therapy with opioids, intake of any analgesic drug within 48 h before surgery.
4. .Subject has Pregnancy, psychiatric disease.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Inability to understand the Study Information Sheet and provide a written consent to take part in the study.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wang Guolin, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
data not entered

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2017 to September 2017, patients were recruited and estimated for eligibility
Pre-assignment Details: Exclusion criteria: coronary heart disease, bronchial asthma, cardiac, lung, hepatic and renal insufficiency, severe hypertension, diabetes mellitus, psychiatric disease, obesity, a history of chronic pain, a history of alcohol or opioid abuse, pregnancy, allergy and contraindication to study drugs.
Groups:
- Dexmedetomidine: Dexmedetomidine is intravenously administrated at a dose of 0.4ug/kg 10min before anesthesia induction until 30min prior to the end of surgery and intraoperative pain management was with remifentanil
  Remifentanil: Remifentanil is intravenously administrated
  Dexmedetomidine: Dexmedetomidine is intravenously administrated before anesthesia induction
- Nalmefene: Nalmefene is intravenously administrated at a dose of 0.3ug/kg before anesthesia induction and intraoperative pain management was with remifentanil
  Remifentanil: Remifentanil is intravenously administrated
  Nalmefene: Nalmefene is intravenously administrated before anesthesia induction
- Dexmedetomidine-Nalmefene: A dose of 0.3ug/kg nalmefene and a dose of 0.4ug/kg dexmedetomidine for 10 minutes before anesthesia induction until 30min prior to the end of surgery and intraoperative pain management was with remifentanil
  Remifentanil: Remifentanil is intravenously administrated
  Dexmedetomidine: Dexmedetomidine is intravenously administrated before anesthesia induction
  Nalmefene: Nalmefene is intravenously administrated before anesthesia induction
Period: Overall Study
Arm/Group | Normal Saline | Sufentanil | Dexmedetomidine | Nalmefene | Dexmedetomidine-Nalmefene
Started | 30 | 30 | 30 | 30 | 30
Completed | 27 | 27 | 27 | 27 | 27
Not Completed | 3 | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine: Dexmedetomidine is intravenously administrated at a dose of 0.5ug/kg 10min before anesthesia induction and intraoperative pain management was with remifentanil
  Remifentanil: Remifentanil is intravenously administrated
  Dexmedetomidine: Dexmedetomidine is intravenously administrated before anesthesia induction
- Dexmedetomidine-Nalmefene: A dose of 0.2ug/kg nalmefene and a dose of 0.5ug/kg dexmedetomidine for 10 minutes before anesthesia induction and intraoperative pain management was with remifentanil
  Remifentanil: Remifentanil is intravenously administrated
  Dexmedetomidine: Dexmedetomidine is intravenously administrated before anesthesia induction
  Nalmefene: Nalmefene is intravenously administrated before anesthesia induction
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Sufentanil | Dexmedetomidine | Nalmefene | Dexmedetomidine-Nalmefene | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (5.0) | 46.0 (8.0) | 45.0 (12) | 47.0 (10) | 46.0 (9) | 46.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 27 | 27 | 27 | 135
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 27 | 27 | 27 | 27 | 27 | 135
Weight [Mean (Standard Deviation); unit: Kg] | 60 (7) | 57 (8) | 59 (7) | 58 (5) | 60 (8) | 59 (7)

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Hyperalgesia Threshold on the Dominant Inner Forearm
Description: The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament at 24 hours postoperatively
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Normal Saline | Sufentanil | Dexmedetomidine | Nalmefene | Dexmedetomidine-Nalmefene
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
g | 61.5 (6.0) | 88.2 (23.40) | 73.0 (3.2) | 67.2 (3.3) | 74.0 (9.3)

2. Secondary Outcome: Normalized Area of Hyperalgesia Around the Incision
Description: The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a 'painful', 'sore' or 'sharper' feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.
Time Frame: 1hours,3hours，6hours，12hours，24hours after surgery
Reporting Status: Not Posted, anticipated posting 2021-12

3. Secondary Outcome: Pain Score (Numerical Rating Scale)
Description: The pain score at rest was evaluated by pain 11-point numerical rating scale : 0 = no pain, 10 = greatest imaginable pain.
Time Frame: 1hours,3hours，6hours，12hours，24hours after surgery
Reporting Status: Not Posted, anticipated posting 2021-12

4. Secondary Outcome: Time of First Postoperative Analgesic Requirement
Description: First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Time Frame: postoperative 1 hours
Reporting Status: Not Posted

5. Secondary Outcome: Cumulative Sufentanyl Consumption
Description: Each patient was administered analgesics using a PCA pump containing sufentanil (100μg) in normal saline at a total volume of 100 ml after leaving post-anaesthesia care unit . This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 24 hours postoperatively
Time Frame: 1hours,3hours，6hours，12hours，24hours after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Occurrence of Side Effects
Description: Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus，hypotention/hypertention，bradycardia/tachycardia
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Incidence of adverse effects was evaluated during 24h after surgery
Arm/Group | Normal Saline | Sufentanil | Dexmedetomidine | Nalmefene | Dexmedetomidine-Nalmefene
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03096730/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03096730/SAP_001.pdf